CLINICAL TRIAL: NCT05752006
Title: Chronic Adaptations to Spinal Flexion Exposure in Crane Operators
Brief Title: Chronic Adaptations to Spinal Flexion Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Matej Voglar, Assistant professor, University of Primorska
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SWE_Flexion2_Crane
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Intervention Model Description: Cross-sectional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crane operators (Experimental): Individuals employed as crane operators in Port of Koper.
  Interventions: Other: Repeated trunk flexion
- Control subjects (Active Comparator): Individuals who spend more than half of their occupation time standing.
  Interventions: Other: Repeated trunk flexion

INTERVENTIONS:
Other: Repeated trunk flexion — A 60-min intermittent trunk flexion protocol. Participants will sit on a standard height sit, with their knees bent at approximately 90° with their hands crossed on their chest. They will perform 40 sets of 60 s of maintaining a flexed position, interspersed with 30 s of rest. Participants will achieve the flexed position by tilting the pelvis posteriorly and leaning forward. During rest, participants will sit up straight without leaning on the support.

SUMMARY:
An experimental study, which will aim to compare changes of trunk mechanical properties and neuromuscular control following spinal flexion exposure in crane operators and control subjects.

DETAILED DESCRIPTION:
Our experimental study will include 40 participants, more specifically 15 crane operators and 15 control subjects. All participants will complete a 60-min protocol of intermittent trunk flexion. Measurements of trunk mechanical properties and neuromuscular control will be performed prior to and following the 60-min protocol.

ELIGIBILITY:
Inclusion Criteria:

* Crane operators: employed as crane operators for more than 3 years
* Occupational workers with a predominantly non static job (e.g. combination of sitting and standing)

Exclusion Criteria:

* History of chronic low back pain
* Episode of acute low back pain
* Hip injury in the past six months
* Previous spine, pelvis or hip surgery
* Hypermobility, diagnosed with the Beighton score
* High intensity resistance training (> 75 % of 1 repetition maximum) more than two times a week
* Control group: sporting or recreational activities, that include repetitive spinal flexion or maintenance of a flexed posture (for example cycling or rowing).

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants will be included, due to gender specificity of crane operators.
Enrollment: 30 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness | 90 minutes
  Muscle stiffness will be measured using ultrasound-based shear wave elastography during prone lying and forward stooping. Erector spinae and multifidus muscle stiffness will be expressed as the shear modulus value in kilopascals.

SECONDARY OUTCOMES:
Change in range of motion | 90 minutes
  Trunk flexion range of motion will be evaluated using Spinal Mouse in maximal trunk flexion while standing.
Change in length of the spine | 90 minutes
  The length of spine will be measured on a custom-developed stadiometer, with the participants in a seated position.
Change in muscle activity | 90 minutes
  Muscle activity will be measured using electromyography during standing, a forward stoop hold and during maximal trunk flexion.
Change in lumbar lordosis angle | 90 minutes
  The lumbar lordosis angle will be evaluated using Spinal Mouse during upright standing.
Change in trunk extension maximal strength | 90 minutes
  Isometric trunk extension peak torque will be assessed on a trunk dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Matej Voglar, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Primorska, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Coded individual data will be uploaded on public scientific data repository.
Supporting Information: Study Protocol